CLINICAL TRIAL: NCT02812953
Title: Biological Collection and Registry of Patients Who Will Have a TAVR (Transcatheter Aortic Valve Replacement) Intervention
Acronym: BIO TAVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Action, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-A01832-47
Record Dates: First submitted 2016-05-30; First posted 2016-06-24 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Platelet poor plasma for von Willebrandt Factor further evaluation
Oversight: Data Monitoring Committee: No

SUMMARY:
A sample of plasma and whole blood will be obtained at 4 time points (pre-procedural, early post-procedural, at hospital discharge and during an eventual visite at 3 or 6 months post-procedural). Test for platelet reactivity (LTA, light transmittance aggregometry and Elisa PRI, Platelet reactivity index), multimeric VWF (von Willebrand factor) and blood level of NET: neutrophil extracellular traps(flow cytometry and ELISA) analyses will be performed at the time of blood sampling. Aliquots of plasma will be stored and frozen for further analyses

DETAILED DESCRIPTION:
There are two major objectives:

* To correlate changes in VWF, platelet reactivity and blood level of NET after TAVR with clinical outcomes
* To correlate changes in VWF, platelet reactivity and blood level of NET with antithrombotic regimens after TAVR (direct anticoagulants apixaban versus standard of care, ie Vitamin K antagonist or antiplatelet therapy).

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing TAVR intervention
* agreement given

Exclusion Criteria:

* severe thrombopenia ( <40.10^9/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing TAVR
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events | 12 months
  stroke/transient ischemic attack; acute coronary syndrome; hospitalization for cardiac insufficiency, cardiovascular or unexplained deaths will be collected at 12 month by phone contact with the patient or his/her relatives or his/her treating physician
Bleeding | 12 months
  Serious bleeding event (BLEED II or more) will be collected at 12 month by phone contact with the patient or his/her relatives or his/her treating physician

SECONDARY OUTCOMES:
mean pressure transprosthetic gradient | within ten days after valve replacement
  value of the mean pressure transprosthetic gradient after TAVR procedure will be assessed by TTE (transthoracic echography) or TOE (transesophageal echography)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pitie Salpetriere, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided